CLINICAL TRIAL: NCT04463628
Title: Impacts of the Covid-19 Epidemic and Associated Lockdown Measures on the Management, Health and Behaviors of Cystic Fibrosis Patients During the 2020 Epidemic
Acronym: MUCONFIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: MUCONFIN
Record Dates: First submitted 2020-06-29; First posted 2020-07-09 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-05

CONDITIONS: Cystic Fibrosis in Children; Cystic Fibrosis
Keywords: Lockdown; Covid-19 Epidemic; questionnaire; interview
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire and/or interview: An online questionnaire to assess the quantitative aspect of the impact of lockdown on all areas of the cystic fibrosis patient's health, be it physical, mental or social (using quality of life assessment in particular and interviews in the human and social sciences).
  Interventions: Behavioral: Questionnaire; Behavioral: Interview

INTERVENTIONS:
Behavioral: Questionnaire — The study questionnaire was constructed as follows:
  * One part is composed of validated questionnaires: Cystic fibrosis specific self-questionnaire for quality of life, questionnaire for screening for anxiety disorder.
  * The other part, which was not validated, was constructed as follows: questionnaire on knowledge of Covid-19 adapted to the new exceptional situation (Covid-19 pandemic) and specific questions adapted to the research objective on Covid-19 from the questionnaire of the French Public Health survey, to monitor changes in behaviour and mental health during lockdown
  Other Names: Quantitative aspect
Behavioral: Interview — Two interviews in the human and social sciences, conducted by recorded video-conference, will be proposed to 15 patients during and after the lockdown.Two interviews will take place: one during the lockdown and one at 6 months from the first interview (or at the end of the confinement if it lasts more than 6 months). The interviews will be conducted independently of the results of the questionnaire.
  Other Names: Qualitative aspect

SUMMARY:
Impacts of the Covid-19 epidemic and associated lockdown measures on the management, health and behaviors of cystic fibrosis patients during the 2020 epidemic

DETAILED DESCRIPTION:
The containment of the population in France is a health measure implemented in response to SARS-CoV-2 (Covid-19) infection. For cystic fibrosis, as for many chronic diseases, this disruption is twofold. On the one hand, it affects daily life due to the closure of schools and the introduction of national lockdown, but also the hospital, which has profoundly changed its procedures, which are almost completely focused on the care of patients with Covid-19. This forced transformation was at the expense of its usual role including the management of chronic diseases such as cystic fibrosis. It has an impact on patients' consultations cancelled, rescheduled or replaced by teleconsultations, hospitalisations whether scheduled or during acute exacerbations which are more complicated to organise. Access to treatments is also more difficult (physiotherapy), which can affect compliance. Confinement also profoundly changes the lives of our patients. It changes the way individuals can apprehend their disease and its integration into their everyday life, studies or professional projects. Finally, it is the confrontation with a potentially fatal infection that reminds us of the risks and consequences of a potentially severe chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cystic fibrosis (Southern Chlorine > 60 mEq/L and/or presence of 2 pathogenic mutations on the CFTR gene)
* Supported in a French CRCM (Cystic fibrosis Resource and Competence Center)
* Affiliated to a social security scheme
* Non-opposition for participation in the protocol

Exclusion Criteria:

* Minor patient under 14 years of age
* Computer equipment or internet connection defect

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be proposed to cystic fibrosis patients residing in France.
Sampling Method: Non-Probability Sample
Enrollment: 746 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Cancellation or postponement of consultations by the health professional or patient, | Up to 6 months
  Number of consultations cancelled or postponed by the health professional or patient of consultations (medical and paramedical),
Patient cancellation of teleconsultations/telecare replacement, | Up to 6 months
  Number of consultations cancelled by the teleconsultation/replacement patient,
Cancellation or postponement by the health care institution or by the patient of hospitalizations (scheduled or unscheduled), | Up to 6 months
  Number of consultations cancelled or postponed by the health care institution or by the patient of hospitalizations (acute or scheduled)
Change in the modalities of administration of antibiotics cures (oral instead of intravenous administration). | Up to 6 months
  Number of patients affected by the change in the modality of administration of antibiotic cures (intravenous instead of intravenous administration).

SECONDARY OUTCOMES:
The reduction of each of the elements of care provision and health care utilization: | Up to 6 months
  Cancellation or postponement by the patient of consultations (medical or paramedical)
  * Patient cancellation of teleconsultations/telecare proposed by the health professional
  * Cancellation or postponement by the patient of hospitalizations (acute or scheduled)
The change of modality of administration of antibiotic cures | Up to 6 months
  Intravenous instead of intravenous administration
Compliance | Up to 6 months
  Questionnaire about taking or not taking treatment during confinement
Anxiety and stress (at risk of being affected by COVID-19 or at risk of being treated less well) | Up to 6 months
  Scale 0-21
Presence or absence of toxic consumption (drug, alcohol) during the lockdown | Up to 6 months
  A questionnaire on the presence or absence of toxic consumption
Evaluation of the knowledge, experience and social representations of the risk of Covid-19 | Up to 6 months
  Experience and social representations of confinement by cystic fibrosis patients (evaluated by qualitative methods)
Assessing the role of social inequalities in the consequences of lockdown | Up to 6 months
  Role of social inequalities in the consequences of containment assessed by qualitative methods
Suspected and/or confirmed Covid-19 in patients with cystic fibrosis. | Up to 6 months
  Prevalence of suspected and/or confirmed Covid-19 infections in patients with cystic fibrosis

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Intercommunal hospital of Créteil, Créteil, IDF
  - TROUSSEAU Hospital, Paris, IDF
  - FOCH Hospital, Suresnes, IDF

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oubaya N, Pombet T, Delestrain C, Remus N, Douvry B, Grenet D, Corvol H, Thouvenin G, Pruliere-Escabasse V, Mounir H, Argoud D, Fretigne C, Costes L, Mackiewicz MP, Jung C, Ahamada L, Lanone S, Maitre B, Begot AC, Epaud R. Impact of the COVID-19 pandemic and associated lockdown measures on the management, health, and behavior of the cystic fibrosis population in France during 2020 (MUCONFIN). Front Public Health. 2022 Nov 14;10:978627. doi: 10.3389/fpubh.2022.978627. eCollection 2022. PMID 36452951